CLINICAL TRIAL: NCT04594304
Title: Screening While You Wait 2: Alcohol and Tobacco Use
Acronym: SWYW2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Women's College Hospital (Other)
Responsible Party: Principal Investigator, Payal Agarwal, Principal Investigator, Women's College Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2019-0002-E
Record Dates: First submitted 2020-06-23; First posted 2020-10-20 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Alcohol; Harmful Use; Tobacco Use; Tobacco Use Cessation; Alcohol Use, Unspecified
MeSH Terms: conditions — Tobacco Use; Tobacco Use Cessation; Alcohol Drinking

STUDY DESIGN:
Intervention Model Description: An independent statistician following a 2:1 ratio to increase opportunities to learn about the intervention processes during this pilot trial will randomly allocate consenting patients following the completion of their baseline survey to intervention or usual care using a computer-generated sequence.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The sequence will be concealed to primary care providers and study staff other than the research coordinator who will apply the allocation. Study staff, including analysts, will also be blind to treatment allocation. Patients and healthcare professionals who may interact with study participants cannot be blinded due to the nature of the intervention, but outcome assessment will be blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized eToolkit (Experimental): The intervention arm will receive a personalized eToolkit with community and electronic supports upon survey completion, and their PCP will receive automatic supports in the EMR to assess and treat the patient's alcohol and/or tobacco use. In cases where a patient does not have risky alcohol and tobacco use, a personalized eToolkit based on their physical activity levels will be administered, and their PCP will receive automatic supports in the EMR to facilitate physical activity discussions. Intervention arm patient participants will be asked to complete a baseline e-survey before their scheduled appointment, a process evaluation e-survey 3 days following their appointment, and a 3 months follow-up e-survey following their appointment. Resources will be automatically produced for the patient and PCP following completion of the baseline e-survey.
  Interventions: Behavioral: Behavioral: Usual care plus eToolkit
- Usual care (No Intervention): The control arm will not receive intervention materials. Control arm patient participants will be asked to complete a baseline e-survey before their scheduled appointment, a process evaluation e-survey 3 days following their appointment, and 3 months follow-up e-survey following their appointment.

INTERVENTIONS:
Behavioral: Behavioral: Usual care plus eToolkit — A baseline e-survey will be sent to participants prior to their scheduled appointment to collect baseline alcohol/tobacco use levels as well as a series of questions evaluating precursors to behaviour change. If randomized into the intervention group, patients will be sent a link to a tailored toolkit based on their behaviours, motivation to change and other pertinent factors. Patients who identify as non-smokers and meet the low-risk drinking guideline, will complete a third screening survey for physical activity. The cumulative patient profile (CPP) status for the patient for alcohol/smoking will be automatically updated post-baseline survey, and the PCP will receive a notification via EMR about the status update. For patients identifying with risky behaviours, the PCP will receive a prompt to update the CPP for the patient and will receive a link, embedded in the EMR, to a PCP-facing toolkit that facilitates evidence-based intervention.
  Arms: Personalized eToolkit

SUMMARY:
This project aims to help patients improve their health through screening and treatment of risky alcohol and tobacco use. Previous studies show the best approach to reduce substance use includes routine screening, short discussions with a clinician, and tailored resources. Unfortunately, primary care providers (PCPs) do not often screen or provide evidence-based interventions. PCPs report lack of confidence, lack of awareness, and competing priorities as barriers to screening and providing evidence-based care. However, digital solutions can enable patient-initiated screening and overcome barriers in a manner that has the potential to be both efficient and effective.

The proposed project will test the feasibility of digital patient-initiated screening at the WCH Family Practice (WCH FP) for alcohol and tobacco use, building on work from the first iteration of Screen While You Wait (SWYW). The research team will email patients a secure link to a survey with screening questions assessing substance use and important contextual factors. The results will be summarized in the patient's chart with an automatic notification to the PCP. If the survey reveals risky behaviours, both the PCP and patient will receive a package of tailored resources for further care delivered through a customized website.

DETAILED DESCRIPTION:
Burden of Alcohol and Tobacco: According to the World Health Organization (WHO), approximately 5.9% of total global deaths are attributable to alcohol consumption. It is estimated that tobacco kills more than 7 million people each year globally. In Ontario alone, approximately 9,800 new cases of cancer diagnosed in a single year could be attributed to tobacco, while 1,000 cases a year could be attributed to alcohol consumption. Despite this evidence, 15.2% of Canadian adults reported drinking more alcohol than the low-risk guidelines, while 15% reported using a tobacco product in the last 30 days.

Addressing Alcohol and Tobacco Together: The health issues associated with tobacco and alcohol use are diverse and pervasive. Many of the health concerns associated with each substance are exacerbated by use of the other (i.e. smokers who also drink alcohol are at an increased risk for cancers of the oral cavity). Further, it has been found that Ontarians who drink alcohol above the recommended safe guidelines are more likely to be smokers. It thus follows that any widespread screening program should target identification of both behaviours. This is supported by recent work that found that alcohol and tobacco use are "often treated separately despite concurrent treatment potentially leading to better outcomes for each".

PCPs are uniquely positioned to impact health behaviours of their patients. Strong evidence and relevant guidelines encourage PCPs to consistently ask about tobacco and alcohol use as a crucial first step to identifying and treating risky behaviours. However, current clinical practice does not live up to these guidelines. A recent report showed that only 23% of patients in Canada had spoken with their providers about alcohol use in the past two years. Furthermore, screening is often limited to periodic health exam visits (i.e. 'complete physicals'), leading to missed opportunities to screen at visit types which may provide key teachable moments, as well as missing patients who may not be coming in for preventative health visits.

Digital, patient-initiated screening is increasingly being recognised as a promising method to improve screening rates by overcoming commonly identified screening barriers. Several small-scale studies have shown that digital, patient-initiated screening can be an efficient method of systematic screening in primary care with high acceptance and usability by patients. These methods may also empower patients to become more engaged in their own health care, particularly those who are both most likely to have risky behaviours and least likely to book preventative care visits.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged >18 who are rostered at WCH FP and have a clinical appointment booked with their PCP in the next 2 weeks
* Have an email address in their EMR chart, and
* Are under-screened for alcohol or tobacco use defined as either a) missing a tobacco or alcohol use status documented in the appropriate section of the cumulative patient profile (CPP) in their EMR or b) having an alcohol or tobacco use status that is positive (defined as any status but: ex-smoker, non-smoker, "rare"-drinker or non-drinker) and no CPX in the last year.

Exclusion Criteria:

* Patients booked for an urgent care appointment (noted in the EMR), as it would not be appropriate to ask patients with acute issues (i.e., short-term severe injury or illness requiring relatively urgent medical attention) to spend extended time receiving alcohol and tobacco use counselling.
* Patients with active risky alcohol or tobacco use who are already undergoing pharmacologic treatment
* Currently pregnant patients will be excluded as pathways for diagnosing, counselling and treating substance use is different among this population. They will be identified through a question before the informed consent form appears asking for the patient's gender. If the patient identifies as a woman, a second question will appear that asks if they are currently pregnant. If yes, the survey will end and the participant will not be asked to complete the consent and survey.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2020-01-02 (Actual); Primary Completion 2021-04-02 (Estimated); Study Completion 2021-08-02 (Estimated)

PRIMARY OUTCOMES:
Updated Cumulative Patient Profile (CPP) Status | Baseline
  Updated CPP statuses for Alcohol and Smoking
Updated Cumulative Patient Profile (CPP) Status | 3 months post appointment
  Updated CPP statuses for Alcohol and Smoking
Discussion around risky substance use in clinic visit | 3 days post appointment
  Patient reported discussion (Y/N) around risky substance use in clinic visit

SECONDARY OUTCOMES:
Level of satisfaction with intervention | 3 days post appointment
  Patient's level of satisfaction (on a 5-point likert scale: Very satisfied, Somewhat satisfied, Neutral, Somewhat dissatisfied, Very dissatisfied) with intervention measured through a process evaluation questionnaire
PCP administration of treatment resources/programs | 3 days post appointment
  Patient reported receival of treatment resources, referrals and programs
PCP administration of treatment resources/programs | 3 months post appointment
  Patient reported receival of treatment resources, referrals and programs
PCP provisioning of pharmacotherapy | 3 days post appointment
  Patient reported receival of prescriptions related to alcohol or tobacco use
PCP provisioning of pharmacotherapy | 3 months post appointment
  Patient reported receival of prescriptions related to alcohol or tobacco use
Patient engagement with personalized toolkit | 3 months post appointment
  Patient reported engagement with toolkit
Patient motivation and self-efficacy to change | Baseline
  Patient self-reported self-efficacy score is determined through 11 questions. Each question is scored from 1-4 (Not at all true, barely true, most true, exactly true). If the participant answers 'mostly true' or 'exactly true' to the majority of the statements (score of 30 or more) they have high self-efficacy. If participant answers 'barely true' or 'not at all true' to the majority of the statements (score of 29 or below), they have low self-efficacy.
Patient motivation and self-efficacy to change | 3 months post appointment
  Patient self-reported self-efficacy score is determined through 11 questions. Each question is scored from 1-4 (Not at all true, barely true, most true, exactly true). If the participant answers 'mostly true' or 'exactly true' to the majority of the statements (score of 30 or more) they have high self-efficacy. If participant answers 'barely true' or 'not at all true' to the majority of the statements (score of 29 or below), they have low self-efficacy.
Patient use of alcohol | Baseline
  Patient reported number of drinks per week. A higher score is likely to indicate harmful drinking or alcohol dependence.
Patient use of alcohol | Baseline
  AUDIT score. A score of 8 or more is associated with harmful or hazardous drinking. A score of 13 or more in women, and 15 or more in men, is likely to indicate alcohol dependence.
Patient use of alcohol | 3 months post appointment
  Patient reported number of drinks per week. A higher score is likely to indicate harmful drinking or alcohol dependence.
Patient use of alcohol | 3 months post appointment
  AUDIT score. AUDIT score. A score of 8 or more is associated with harmful or hazardous drinking. A score of 13 or more in women, and 15 or more in men, is likely to indicate alcohol dependence.
Patient use of tobacco | Baseline
  Patient reported number of cigarettes per week. A higher number is likely to indicate increased risk for negative health outcomes.
Patient use of tobacco | 3 months post appointment
  Patient reported number of cigarettes per week. A higher number is likely to indicate increased risk for negative health outcomes.
Proportion of consent | Baseline
  Proportion of patients that consented, completed the surveys at each time interval, and at follow-up (with reasons for refusal if applicable)
Proportion of consent | 3 days post appointment
  Proportion of patients that consented, completed the surveys at each time interval, and at follow-up (with reasons for refusal if applicable)
Proportion of consent | 3 months post appointment
  Proportion of patients that consented, completed the surveys at each time interval, and at follow-up (with reasons for refusal if applicable)

CONTACTS AND LOCATIONS:
Overall Officials: Payal Agarwal, MD, Principal Investigator — Women's College Hospital
Locations (1):
- Women's College Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Minian N, Baliunas D, Zawertailo L, Noormohamed A, Giesbrecht N, Hendershot CS, Le Foll B, Rehm J, Samokhvalov A, Selby PL. Combining alcohol interventions with tobacco addictions treatment in primary care-the COMBAT study: a pragmatic cluster randomized trial. Implement Sci. 2017 May 18;12(1):65. doi: 10.1186/s13012-017-0595-7. PMID 28521782
- [Background] Papadakis S, Cole AG, Reid RD, Coja M, Aitken D, Mullen KA, Gharib M, Pipe AL. Increasing Rates of Tobacco Treatment Delivery in Primary Care Practice: Evaluation of the Ottawa Model for Smoking Cessation. Ann Fam Med. 2016 May;14(3):235-43. doi: 10.1370/afm.1909. PMID 27184994
- [Background] Carey M, Noble N, Mansfield E, Waller A, Henskens F, Sanson-Fisher R. The Role of eHealth in Optimizing Preventive Care in the Primary Care Setting. J Med Internet Res. 2015 May 22;17(5):e126. doi: 10.2196/jmir.3817. PMID 26001983
- [Background] Kumar PC, Cleland CM, Gourevitch MN, Rotrosen J, Strauss S, Russell L, McNeely J. Accuracy of the Audio Computer Assisted Self Interview version of the Alcohol, Smoking and Substance Involvement Screening Test (ACASI ASSIST) for identifying unhealthy substance use and substance use disorders in primary care patients. Drug Alcohol Depend. 2016 Aug 1;165:38-44. doi: 10.1016/j.drugalcdep.2016.05.030. Epub 2016 Jun 22. PMID 27344194
- [Background] Rogausch A, Sigle J, Seibert A, Thuring S, Kochen MM, Himmel W. Feasibility and acceptance of electronic quality of life assessment in general practice: an implementation study. Health Qual Life Outcomes. 2009 Jun 3;7:51. doi: 10.1186/1477-7525-7-51. PMID 19493355
- [Background] Hess R, Santucci A, McTigue K, Fischer G, Kapoor W. Patient difficulty using tablet computers to screen in primary care. J Gen Intern Med. 2008 Apr;23(4):476-80. doi: 10.1007/s11606-007-0500-1. PMID 18373148